CLINICAL TRIAL: NCT06179732
Title: Field Evaluations of Innovative Tools for Vector-borne Disease Control in Conflict-affected Communities:A Cluster Randomised Trial
Brief Title: Field Evaluations of Innovative Tools for Vector-borne Disease Control in Conflict-affected Communities
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Mentor Initiative (Other)
Collaborators: Liverpool School of Tropical Medicine (Other); University of Maiduguri (Other); US government (Unknown); SCJohnson (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USDA01YEM - Nigeria
Record Dates: First submitted 2023-11-10; First posted 2023-12-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-06

CONDITIONS: Malaria; Childhood ALL; Vector Borne Diseases
Keywords: malaria; cluster randomised trial; children; vector borne diseases; Nigeria; Internally Displaced People camps
MeSH Terms: conditions — Malaria; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Vector Borne Diseases | interventions — transfluthrin

STUDY DESIGN:
Masking Description: Neither the deliverers of the intervention nor the outcome assessors are blinded to the group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): 1. Information and Education Campaigns (IEC) campaigns will formally encourage breeding site management through; good practice household-level water storage (covering and cleaning of water storage containers) and waste management (removal of potential breeding sites in and around the home).
  2. Epidemiological surveillance: test and treat malaria cases in children 6 - 10 years of age
- Mesh (Experimental): 1. Information and Education Campaigns (IEC) campaigns will formally encourage breeding site management through; good practice household-level water storage (covering and cleaning of water storage containers) and waste management (removal of potential breeding sites in and around the home).
  2. Epidemiological surveillance: test and treat malaria cases in children 6 - 10 years of age
  3. Mesh product distributed to households
  Interventions: Combination Product: Mesh - spatial repellent impregnated with transfluthrin (2500mg); Behavioral: Information and Education Campaigns (IEC); Diagnostic Test: test and treat malaria cases

INTERVENTIONS:
Combination Product: Mesh - spatial repellent impregnated with transfluthrin (2500mg) — Mesh is one of the first spatial repellent tools to provide long-lasting protection to users, with predicted efficacy of 6-months. The active ingredient of Mesh is transfluthrin, a fast-acting volatile pyrethroid with low persistency, which can act either by killing or via sublethal toxicity that causes deviation (repellency) in host attraction, reducing host-contact and risk of infectious bites. The chemical passively releases into the air and interacts with vector odour receptors causing irritation. The design of Mesh is simple with a transfluthrin-infused sheet protected by plastic mesh and encased in a plastic frame.
  Mesh will be distributed to the intervention arm only.
  Arms: Mesh
Behavioral: Information and Education Campaigns (IEC) — IEC campaigns will formally encourage breeding site management through; good practice household-level water storage (covering and cleaning of water storage containers) and waste management (removal of potential breeding sites in and around the home) using leaflets and word of mouth. IEC will be conducted in both arms.
  Arms: Mesh
Diagnostic Test: test and treat malaria cases — All children in the cohort (both arms) will be tested by rapid diagnostic testing (RDT) monthly. If any children test positive, they will be treated with a course of 3-day artemisinin combination therapy (ACT) according to standard protocol and local guidelines. All children in the cohort will receive ACT to provide clearance of any malaria parasites during the baseline of the study.
  Arms: Mesh

SUMMARY:
The aim of this study is to determine the effectiveness of a new spatial repellent (called Mesh) at repelling multiple disease vectors and, reducing clinical malaria rates in temporary shelters and camp settings. The design of the study will be a two-armed cluster randomised trial.

By conducting the research in challenging camp settings in the north of Nigeria, the MENTOR Initiative aims to determine whether Mesh can be effective in harsh camp conditions where communities are living in conflict area temporary shelters.

ELIGIBILITY:
Inclusion Criteria:

* Shelters with 1 or more children from 6-10 years old
* Shelters with an adult/head of the household

Exclusion Criteria:

* Shelters without children from 6-10 years old

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
entomological outcome: vector density | 7 months
  the relative infestation rate of disease vectors (females of any of Anopheles malaria vectors, Aedes aegypti, or phlebotomine sand flies
epidemiological outcome: malaria incidence | 7 months
  Malaria incidence will be estimated as the total number of malaria episodes per person over the course of the trial.

SECONDARY OUTCOMES:
feasibility, acceptance and uptake of Mesh | 7 months
  To measure community and household acceptance and uptake of Mesh, a questionnaire will be conducted with the Mesh-receiving households.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Allan, Principal Investigator — The Mentor Initiative
Locations (1):
- Sara Estecha Querol, Haywards Heath, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allan RJ, Scherrer R, Estecha-Querol S, Weetman D, Paris L, Ba'abba Goni U, Idris Abdulhamid F, Nfornuh Alenwi B, Ahmad S, Cross CL, Ashir GM, Waziri M, Ntadom G, Messenger LA. The effectiveness of long-lasting spatial repellent emanators against malaria in humanitarian crisis settings in northern Nigeria: a two-arm pragmatic, open-label, controlled trial. Lancet Infect Dis. 2026 Jan 8:S1473-3099(25)00684-X. doi: 10.1016/S1473-3099(25)00684-X. Online ahead of print. PMID 41520670